CLINICAL TRIAL: NCT04911920
Title: Validation of a German Version of the Patient Rated Tennis Elbow Evaluation (PRTEE)
Brief Title: Validation of a German Version of the Patient Rated Tennis Elbow Evaluation
Acronym: PRTEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miriam Marks (Other)
Responsible Party: Sponsor-Investigator, Miriam Marks, Research Associate, Schulthess Klinik
Organization: Schulthess Klinik (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OE-0141
Record Dates: First submitted 2021-05-21; First posted 2021-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Elbow Tendinitis; Elbow, Tennis
Keywords: Questionnaire; PRTEE
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with lateral epicondylitis (Other): Patients with lateral epicondylitis who are treated with at least one ACP injection.
  Interventions: Other: Questionnaire Patient Rated Tennis Elbow Evaluation

INTERVENTIONS:
Other: Questionnaire Patient Rated Tennis Elbow Evaluation — Participants are asked to complete questionnaires at three measurement time points.

SUMMARY:
The German version of the Patient Rated Tennis Elbow Evaluation (PRTEE) questionnaire is tested for reliability, validity and responsiveness.

DETAILED DESCRIPTION:
In this prospective study, patients with lateral epicondylitis will complete the PRTEE before ACP injection, 6 weeks after treatment and 2-11 days later.

The statistics will include analyses about reliability, validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosed lateral epicondylitis
* Receive a first ACP treatment at the Schulthess Klinik
* Signed informed consent form

Exclusion Criteria:

* Lack of German language skills, which make it impossible to complete the questionnaire
* Diseases or conditions that would prevent accurate evaluation (e.g. central neurological, psychiatric or metabolic diseases)
* Legal incompetence
* Recent operations on the elbow or hand (less than three months ago)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire Patient Rated Tennis Elbow Evaluation | Ten Weeks
  Participants are asked to complete questionnaires at each of three measurement time points.

SECONDARY OUTCOMES:
Sociodemographic data | Ten Weeks
  The socio-demographic data includes the patient's age, sex, duration of symptoms, handedness and disease-related data
The Disabilities of Arm Shoulder and Hand (DASH) questionnaire | Ten Weeks
  The patient questionnaire measures impairment of the upper extremity
The Patient Rated Elbow Evaluation (PREE) | Ten Weeks
  It measures the elbow specific pain and limitations
EQ-5D-5L | Ten Weeks
  general measure of health for clinical and economic questions
Patient satisfaction Questionnaire | Ten Weeks
  perceived change regarding their elbow condition

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Marks, PhD, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No